CLINICAL TRIAL: NCT03545217
Title: Abnormal Glucose Metabolism in HIV-infected Patients: Prevalence of Prediabetes, the Relationship to Gut Microbiota and Sleep, and the Role of Lifestyle Intervention
Brief Title: Abnormal Glucose Metabolism in HIV-infected Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Somnuek Sungkanuparph, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID066011
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Abnormal Glucose Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: Lifestyle Intervention
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle Intervention — a 6-month intensive lifestyle intervention program led by a multidisciplinary team of diabetes nurses and dieticians, and a follow up at 12 months for these participants. This will be a group-based activity adapted from the Diabetes Prevention Program -Thailand project
  Arms: intervention group

SUMMARY:
HIV is a major health problem worldwide especially in low-to middle-income countries including Thailand. Fortunately, a significant reduction in morbidity and mortality has been observed due to the use of combination antiretroviral therapy. As the natural history of the disease is modified, non-communicable diseases are becoming recognized complications of HIV infection, including insulin resistance, dyslipidemia and type 2 diabetes. The prevalence of type 2 diabetes in HIV-infected patients is significantly higher than in the general population, likely contributed by antiretroviral regimen and an ongoing, usually subclinical, inflammation. People with prediabetes, a condition which blood sugars are elevated but not yet meeting the criteria for diabetes, represent a high risk group for future diabetes development. Lifestyle interventions, including diet and exercise, are effective in reducing the future diabetes risk by as much as 58%, including in Thailand. The knowledge whether these interventions are effective in HIV-infected patients, given their unique characteristics, is not available at this time but urgently needed. Moreover, the program tailored to each country's local values, culture and socioeconomic status is essential as participants' acceptability is one of the keys to program's success. This current proposal will adapt a 6-month intensive lifestyle intervention program and evaluate its feasibility and acceptability in HIV-infected individuals with prediabetes in Thailand. The knowledge gained will be highly relevant for Thailand and for other low-to-middle-income countries. Furthermore, gut microbiota and insufficient sleep are novel factors shown to affect individual's metabolic health. Insufficient sleep is recognized as a risk factor for incident diabetes. Gut microbiota composition differs between those with and without diabetes. The current proposal will examine how gut microbiota and sleep duration differ between HIV-infected individuals with and without prediabetes, and now there change or modulate the metabolic response to the 6-month intensive lifestyle interventions. Lastly, HIV and diabetes are global epidemics, research capacity building among countries is essential to battle these health problems. This proposal will aim to build research capacities among three international institutions: University of Illinois at Chicago, Illinois, U.S.A.; Faculty of Medicine Ramathibodi Hospital, Mahidol University, Thailand, one of the top medical schools in Thailand; and a newly formed medical school, Navamindradhiraj University, Vajira Hospital, Bangkok, Thailand. Through close collaboration, networking, in-person training and workshops, the proposed study will enhance research capacity and improve lives of those living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients, age 35-65 years old
* Receiving antiretroviral therapy
* Diagnosis of prediabetes (hemoglobin A1c, HbA1c levels ≥5.7-<6.5% and fasting glucose levels <126 mg/dl and 2-hour glucose levels <200 mg/dl following 75-gram OGTT)

Exclusion Criteria:

* Serious medical problems (stroke with significant disability, estimated glomerular filtration rate <45 ml/min/1.73 m2, uncontrolled congestive heart failure, symptoms suggestive of untreated cardiopulmonary disease such as chest pain or shortness of breath, significant anemia defined as hemoglobin <9.0 g/dL, severe pulmonary disease including those requiring home oxygen therapy, end stage liver disease)
* A previous diagnosis of diabetes
* Currently diagnosed with contagious infectious disease
* Pregnancy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
new diabetes | 12 months after intervention
  occurrence of diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Somnuek Sungkanuparph, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nimitphong H, Sungkanuparph S, Areevut C, Saetung S, Jerawatana R, Hathaidechadusadee A, Somwang S, Tongchom W, Saibuathong N, Sakmanarit J, Pichitchaipitak O, Phuphuakrat A, Reutrakul S. Effects of an intensive lifestyle intervention and the role of sleep in people living with HIV and prediabetes: a pilot and feasibility study. BMC Res Notes. 2021 Apr 17;14(1):145. doi: 10.1186/s13104-021-05558-z. PMID 33865450
- [Derived] Phuphuakrat A, Nimitphong H, Reutrakul S, Sungkanuparph S. Prediabetes among HIV-infected individuals receiving antiretroviral therapy: prevalence, diagnostic tests, and associated factors. AIDS Res Ther. 2020 May 24;17(1):25. doi: 10.1186/s12981-020-00284-1. PMID 32448349